CLINICAL TRIAL: NCT00934089
Title: A Phase 2, Single-masked, Randomized, Crossover Study Of The 24-hour Intraocular Pressure Lowering And Systemic Exposure of Pf-04217329 Alone And In Combination With Latanoprost
Brief Title: A Phase 2 Study Of The 24-Hour Intraocular Pressure Lowering And Systemic Exposure Of PF-04217329
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: A0191002
Record Dates: First submitted 2009-07-06; First posted 2009-07-08 (Estimated); Results first posted 2021-05-03 (Actual); Last update posted 2021-05-03 (Actual); Status verified 2021-04

CONDITIONS: Glaucoma, Open-Angle; Ocular Hypertension
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension | interventions — PF 04217329; Latanoprost

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- PF-04217329 + placebo (Experimental): Active study drug + latanoprost vehicle
  Interventions: Drug: PF-04217329; Drug: latanoprost vehicle
- PF-04217329 + latanoprost (Experimental): Active study drug + latanoprost
  Interventions: Drug: PF-04217329; Drug: latanoprost

INTERVENTIONS:
Drug: PF-04217329 — Topical ocular solution, once-daily for 14 days
  Arms: PF-04217329 + placebo
Drug: latanoprost vehicle — Topical ocular solution, once-daily for 14 days
  Arms: PF-04217329 + placebo
Drug: PF-04217329 — Topical ocular solution, once-daily for 14 days
  Arms: PF-04217329 + latanoprost
Drug: latanoprost — Topical ocular solution, once-daily for 14 days
  Other Names: Xalatan
  Arms: PF-04217329 + latanoprost

SUMMARY:
This study will characterize the effect of PF-04217329, alone and in combination with latanoprost, on circadian intraocular pressure and blood pressure in glaucoma patients. Blood samples will be collected to measure the amount of active metabolite of PF-04217329 in the plasma following dosing.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of primary open-angle glaucoma or ocular hypertension in one or both eyes
* Intraocular Pressure (IOP) of at least 22 mmHg and not more than 30 mmHg in either eye at 8 AM after discontinuing previous glaucoma treatment
* Visual acuity correctable to 20/100 or better in each eye.

Exclusion Criteria:

* Closed/barely open anterior chamber angle or a history of acute angle closure in either eye.
* Diagnosis of a clinically significant or progressive retinal disease (eg, diabetic retinopathy, macular degeneration) in either eye.
* Advanced glaucoma or a history of severe central visual field loss in either eye.
* History of ocular surgery or trauma in either eye within 6 months of the screening visit.
* History of ocular infection, ocular inflammation, or laser surgery in either eye within 3 months of the screening visit.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2010-01; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (8):
- United States (8):
  - West Coast Clinical Trials, LLC, Cypress, California
  - Glory Medical Group, Garden Grove, California
  - East-West Eye Institute, Gardena, California
  - Ophthalmology Corporation, Long Beach, California
  - East-West Eye Institute, Los Angeles, California
  - Los Angeles Eye Medical Group, Los Angeles, California
  - Eye Research Foundation, Newport Beach, California
  - Southern California Glaucoma Consultants, Pasadena, California

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A0191002&StudyName=A%20Phase%202%20Study%20Of%20The%2024-Hour%20Intraocular%20Pressure%20Lowering%20And%20Systemic%20Exposure%20Of%20PF-04217329

RESULTS

PARTICIPANT FLOW:
Groups:
- Taprenepag+Latanoprost, Then Taprenepag+Latanoprost Vehicle: Participants self-administered 1 drop (27 microliter [mcL]) of latanoprost 0.005 percent (%) ophthalmic solution followed by taprenepag (taprenepag isopropyl, PF-04217329) 0.01% ophthalmic solution into each eye once daily for 14 days in first intervention period and then vehicle matched to latanoprost ophthalmic solution followed by taprenepag (taprenepag isopropyl, PF-04217329) 0.01% ophthalmic solution into each eye once daily for 14 days in second intervention period. A 28-day washout period was maintained between each period.
- Taprenepag+Latanoprost Vehicle,Then Taprenepag+Latanoprost: Participants self-administered 1 drop (27 mcL) of vehicle matched to latanoprost ophthalmic solution followed by taprenepag (taprenepag isopropyl, PF-04217329) 0.01% ophthalmic solution into each eye once daily for 14 days in first intervention period and then latanoprost 0.005% ophthalmic solution followed by taprenepag (taprenepag isopropyl, PF-04217329) 0.01% ophthalmic solution into each eye once daily for 14 days in second intervention period. A 28-day washout period was maintained between each period.
Period: First Intervention Period (14 Days)
Arm/Group | Taprenepag+Latanoprost, Then Taprenepag+Latanoprost Vehicle | Taprenepag+Latanoprost Vehicle,Then Taprenepag+Latanoprost
Started | 15 | 16
Treated | 14 | 16
Completed | 13 | 16
Not Completed | 2 | 0
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Randomized, but not treated | 1 | 0
Period: Washout Period (28 Days)
Arm/Group | Taprenepag+Latanoprost, Then Taprenepag+Latanoprost Vehicle | Taprenepag+Latanoprost Vehicle,Then Taprenepag+Latanoprost
Started | 13 | 16
Completed | 13 | 16
Not Completed | 0 | 0
Period: Second Intervention Period (14 Days)
Arm/Group | Taprenepag+Latanoprost, Then Taprenepag+Latanoprost Vehicle | Taprenepag+Latanoprost Vehicle,Then Taprenepag+Latanoprost
Started | 13 | 16
Completed | 13 | 16
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population included all randomized participants who received at least 1 dose of study medication.
Groups:
- Total: Total of all reporting groups
Arm/Group | Taprenepag+Latanoprost, Then Taprenepag+Latanoprost Vehicle | Taprenepag+Latanoprost Vehicle,Then Taprenepag+Latanoprost | Total
Number analyzed (Participants) | 14 | 16 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.2 (9.0) | 65.2 (11.3) | 66.6 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 11 | 22
  Male | 3 | 5 | 8

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Mean Intra Ocular Pressure (IOP) in Study Eye at Day 14: 8 Ante Meridiem (AM) (0 Hour)
Description: IOP was measured using Perkins applanation tonometer at Day -8, Day 14 and using standard Goldmann applanation tonometer at eligibility visit. IOP was measured in both eyes, and the eye with higher IOP reading across eligibility visit and Day -8 visit was referred as 'study eye' for efficacy assessment. If both measurements were equal, right eye was selected as study eye. IOP was measured twice in same eye, and if difference between 2 measurements was less than or equal to 2 millimeter of mercury (mmHg), mean of the 2 readings was recorded as the IOP at that time point. If the difference between 2 readings was greater than 2 mmHg, a third consecutive reading was taken and the median IOP was recorded as the IOP at that time point. Mean IOP was reported as the average of individual participants' mean or median IOP values. Change from baseline in IOP = baseline IOP - post-baseline IOP. Change was calculated using the value at 8 AM on Day -8 as baseline for 8 AM value on Day 14.
Time Frame: 8 AM on Baseline (Day -8), 8 AM on Day 14 (0 Hour)
Population: Per-protocol (PP) population included all participants who completed the study treatment with no major protocol violations.
Measure: Mean (Standard Deviation); unit: mmHg
Groups:
- Taprenepag+Latanoprost: Participants self-administered 1 drop (27 mcL) of latanoprost 0.005 percent (%) ophthalmic solution followed by taprenepag (taprenepag isopropyl, PF-04217329) 0.01% ophthalmic solution into each eye once daily for 14 days in either first intervention period or second intervention period.
- Taprenepag+Latanoprost Vehicle: Participants self-administered 1 drop (27 mcL) of vehicle matched to latanoprost ophthalmic solution followed by taprenepag (taprenepag isopropyl, PF-04217329) 0.01% ophthalmic solution into each eye once daily for 14 days in either first intervention period or second intervention period.
Arm/Group | Taprenepag+Latanoprost | Taprenepag+Latanoprost Vehicle
Number analyzed (Participants) | 24 | 28
mmHg
  Baseline (Day -8) : 8 AM | 22.77 (3.264) | 22.41 (2.786)
  Change at Day 14: 8 AM | 5.00 (2.391) | 3.79 (2.942)

2. Primary Outcome: Change From Baseline in Mean Intra Ocular Pressure (IOP) in Study Eye at Day 14: 10 AM (2 Hours)
Description: IOP was measured using Perkins applanation tonometer at Day -8, Day 14 and using standard Goldmann applanation tonometer at eligibility visit. IOP was measured in both eyes, and the eye with higher IOP reading across eligibility visit and Day -8 visit was referred as 'study eye' for efficacy assessment. If both measurements were equal, right eye was selected as study eye. IOP was measured twice in same eye, and if difference between 2 measurements was less than or equal to 2 millimeter of mercury, mean of the 2 readings was recorded as the IOP at that time point. If the difference between 2 readings was greater than 2 mmHg, a third consecutive reading was taken and the median IOP was recorded as the IOP at that time point. Mean IOP was reported as the average of individual participants' mean or median IOP values. Change from baseline in IOP = baseline IOP - post-baseline IOP. Change was calculated using the value at 10 AM on Day -8 as baseline for 10 AM value on Day 14.
Time Frame: 10 AM on Baseline (Day -8), 10 AM on Day 14 (2 Hours)
Population: PP population included all participants who completed the study treatment with no major protocol violations.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Taprenepag+Latanoprost | Taprenepag+Latanoprost Vehicle
Number analyzed (Participants) | 24 | 28
mmHg
  Baseline (Day -8): 10 AM | 21.40 (3.022) | 20.82 (2.385)
  Change at Day 14: 10 AM | 3.90 (2.445) | 3.09 (2.822)

3. Primary Outcome: Change From Baseline in Mean Intra Ocular Pressure (IOP) in Study Eye at Day 14: 12 Post Meridiem (PM) (4 Hours)
Description: IOP was measured using Perkins applanation tonometer at Day -8, Day 14 and using standard Goldmann applanation tonometer at eligibility visit. IOP was measured in both eyes, and the eye with higher IOP reading across eligibility visit and Day -8 visit was referred as 'study eye' for efficacy assessment. If both measurements were equal, right eye was selected as study eye. IOP was measured twice in the same eye, and if difference between 2 measurements was less than or equal to 2 millimeter of mercury (mmHg), mean of 2 readings was recorded as IOP at that time point. If the difference between 2 readings was greater than 2 mmHg, a third consecutive reading was taken and the median IOP was recorded as the IOP at that time point. Mean IOP was reported as the average of individual participants' mean or median IOP values. Change from baseline in IOP = baseline IOP - post-baseline IOP. Change was calculated using the value at 12 PM on Day -8 as baseline for 12 PM value on Day 14.
Time Frame: 12 PM on Baseline (Day -8), 12 PM on Day 14 (4 Hours)
Population: PP population included all participants who completed the study treatment with no major protocol violations.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Taprenepag+Latanoprost | Taprenepag+Latanoprost Vehicle
Number analyzed (Participants) | 24 | 28
mmHg
  Baseline (Day -8): 12 PM | 21.54 (3.514) | 21.45 (2.518)
  Change at Day 14: 12 PM | 5.15 (2.482) | 4.43 (2.530)

4. Primary Outcome: Change From Baseline in Mean Intra Ocular Pressure (IOP) in Study Eye at Day 14: 2 PM (6 Hours)
Description: IOP was measured using Perkins applanation tonometer at Day -8, Day 14 and using standard Goldmann applanation tonometer at eligibility visit. IOP was measured in both eyes, and the eye with higher IOP reading across eligibility visit and Day -8 visit was referred as 'study eye' for efficacy assessment. If both measurements were equal, right eye was selected as study eye. IOP was measured twice in same eye, and if difference between 2 measurements was less than or equal to 2 millimeter of mercury (mmHg), mean of the 2 readings was recorded as the IOP at that time point. If the difference between 2 readings was greater than 2 mmHg, a third consecutive reading was taken and the median IOP was recorded as the IOP at that time point. Mean IOP was reported as the average of individual participants' mean or median IOP values. Change from baseline in IOP = baseline IOP - post-baseline IOP. Change was calculated using the value at 2 PM on Day -8 as baseline for 2 PM value on Day 14.
Time Frame: 2 PM on Baseline (Day -8), 2 PM on Day 14 (6 Hours)
Population: PP population included all participants who completed the study treatment with no major protocol violations. Here 'number analyzed' signifies those participants who were evaluable for this measure at given time points for each group, respectively.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Taprenepag+Latanoprost | Taprenepag+Latanoprost Vehicle
Number analyzed (Participants) | 24 | 28
mmHg
  Baseline (Day -8): 2 PM | 22.25 (2.766) | 20.80 (2.601)
  Change at Day 14: 2 PM: number analyzed (Participants) | 24 | 27
  Change at Day 14: 2 PM | 6.56 (2.438) | 3.91 (2.500)

5. Primary Outcome: Change From Baseline in Mean Intra Ocular Pressure (IOP) in Study Eye at Day 14: 4 PM (8 Hours)
Description: IOP was measured using Perkins applanation tonometer at Day -8, Day 14 and using standard Goldmann applanation tonometer at eligibility visit. IOP was measured in both eyes, and the eye with higher IOP reading across eligibility visit and Day -8 visit was referred as 'study eye' for efficacy assessment. If both measurements were equal, right eye was selected as study eye. IOP was measured twice in same eye, and if difference between 2 measurements was less than or equal to 2 millimeter of mercury (mmHg), mean of the 2 readings was recorded as the IOP at that time point. If the difference between 2 readings was greater than 2 mmHg, a third consecutive reading was taken and the median IOP was recorded as the IOP at that time point. Mean IOP was reported as the average of individual participants' mean or median IOP values. Change from baseline in IOP = baseline IOP - post-baseline IOP. Change was calculated using the value at 4 PM on Day -8 as baseline for 4 PM value on Day 14.
Time Frame: 4 PM on Baseline (Day -8), 4 PM on Day 14 (8 Hours)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Taprenepag+Latanoprost | Taprenepag+Latanoprost Vehicle
Number analyzed (Participants) | 24 | 28
mmHg
  Baseline (Day -8): 4 PM | 18.56 (3.383) | 17.68 (3.403)
  Change at Day 14: 4 PM: number analyzed (Participants) | 24 | 27
  Change at Day 14: 4 PM | 5.79 (3.333) | 4.50 (3.611)

6. Primary Outcome: Change From Baseline in Mean Intra Ocular Pressure (IOP) in Study Eye at Day 14: 6 PM (10 Hours)
Description: IOP was measured using Perkins applanation tonometer at Day -8, Day 14 and using standard Goldmann applanation tonometer at eligibility visit. IOP was measured in both eyes, and the eye with higher IOP reading across eligibility visit and Day -8 visit was referred as 'study eye' for efficacy assessment. If both measurements were equal, right eye was selected as study eye. IOP was measured twice in same eye, and if difference between 2 measurements was less than or equal to 2 millimeter of mercury (mmHg), mean of the 2 readings was recorded as the IOP at that time point. If the difference between 2 readings was greater than 2 mmHg, a third consecutive reading was taken and the median IOP was recorded as the IOP at that time point. Mean IOP was reported as the average of individual participants' mean or median IOP values. Change from baseline in IOP = baseline IOP - post-baseline IOP. Change was calculated using the value at 6 PM on Day -8 as baseline for 6 PM value on Day 14.
Time Frame: 6 PM on Baseline (Day -8), 6 PM on Day 14 (10 Hours)
Population: PP population included all participants who completed the study treatment with no major protocol violations.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Taprenepag+Latanoprost | Taprenepag+Latanoprost Vehicle
Number analyzed (Participants) | 24 | 28
mmHg
  Baseline (Day -8): 6 PM | 19.10 (3.369) | 17.29 (3.326)
  Change at Day 14: 6 PM | 6.42 (4.655) | 3.95 (3.417)

7. Primary Outcome: Change From Baseline in Mean Intra Ocular Pressure (IOP) in Study Eye at Day 14: 8 PM (12 Hours)
Description: IOP was measured using Perkins applanation tonometer at Day -8, Day 14 and using standard Goldmann applanation tonometer at eligibility visit. IOP was measured in both the eyes, and eye with higher IOP reading across eligibility visit and Day -8 visit was referred as 'study eye' for efficacy assessment. If both measurements were equal, right eye was selected as study eye. IOP was measured twice in same eye, and if difference between 2 measurements was less than or equal to 2 millimeter of mercury (mmHg), mean of the 2 readings was recorded as the IOP at that time point. If the difference between 2 readings was greater than 2 mmHg, a third consecutive reading was taken and the median IOP was recorded as the IOP at that time point. Mean IOP was reported as the average of individual participants' mean or median IOP values. Change from baseline in IOP = baseline IOP - post-baseline IOP. Change was calculated using the value at 8 PM on Day -8 as baseline for 8 PM value on Day 14.
Time Frame: 8 PM on Baseline (Day -8), 8 PM on Day 14 (12 Hours)
Population: PP population included all participants who completed the study treatment with no major protocol violations.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Taprenepag+Latanoprost | Taprenepag+Latanoprost Vehicle
Number analyzed (Participants) | 24 | 28
mmHg
  Baseline (Day -8) for Day 14 : 8 PM | 18.58 (3.790) | 16.66 (3.483)
  Change at Day 14: 8 PM | 6.44 (4.220) | 3.30 (3.425)

8. Primary Outcome: Change From Baseline in Mean Intra Ocular Pressure (IOP) in Study Eye at Day 14: 10 PM (14 Hours)
Description: IOP was measured using Perkins applanation tonometer at Day -8, Day 14 and using standard Goldmann applanation tonometer at eligibility visit. IOP was measured in both eyes, and the eye with higher IOP reading across eligibility visit and Day -8 visit was referred as 'study eye' for efficacy assessment. If both measurements were equal, right eye was selected as study eye. IOP was measured twice in the same eye, and if difference between 2 measurements was less than or equal to 2 millimeter of mercury (mmHg), mean of 2 readings was recorded as the IOP at that time point. If the difference between 2 readings was greater than 2 mmHg, a third consecutive reading was taken and the median IOP was recorded as the IOP at that time point. Mean IOP was reported as the average of individual participants' mean or median IOP values. Change from baseline in IOP = baseline IOP - post-baseline IOP. Change was calculated using the value at 10 PM on Day -8 as baseline for 10 PM value on Day 14.
Time Frame: 10 PM on Day -8 (Baseline), 10 PM on Day 14 (14 Hours)
Population: PP population included all participants who completed the study treatment with no major protocol violations.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Taprenepag+Latanoprost | Taprenepag+Latanoprost Vehicle
Number analyzed (Participants) | 24 | 28
mmHg
  Baseline (Day -8): 10 PM | 18.25 (2.978) | 17.96 (3.347)
  Change at Day 14: 10 PM | 5.40 (3.365) | 3.88 (3.693)

9. Primary Outcome: Change From Baseline in Mean Intra Ocular Pressure (IOP) in Study Eye at Day 15: 12 AM (16 Hours)
Description: IOP was measured using Perkins applanation tonometer at Day -8 and using standard Goldmann applanation tonometer at eligibility visit, Day -7 and Day 15. IOP was measured in both eyes, and the eye with higher IOP reading across eligibility visit and Day -8 was referred as 'study eye' for efficacy assessment. If both measurements were equal, right eye was selected as study eye. IOP was measured twice in the same eye, and if difference between 2 measurements was less than or equal to 2 millimeter of mercury (mmHg), mean of 2 readings was recorded as IOP at that time point. If the difference between 2 readings was greater than 2 mmHg, a third consecutive reading was taken and the median IOP was recorded as the IOP at that time point. Mean IOP was reported as the average of individual participants' mean or median IOP values. Change from baseline in IOP = baseline IOP - post-baseline IOP. Change was calculated using the value at 12 AM on Day -7 as baseline for 12 AM value on Day 15.
Time Frame: 12 AM on Baseline (Day -7), 12 AM on Day 15 (16 Hours)
Population: PP population included all participants who completed the study treatment with no major protocol violations.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Taprenepag+Latanoprost | Taprenepag+Latanoprost Vehicle
Number analyzed (Participants) | 24 | 28
mmHg
  Baseline (Day -7): 12 AM | 17.98 (3.580) | 16.77 (3.770)
  Change at Day 15: 12 AM | 5.71 (2.400) | 4.34 (3.443)

10. Primary Outcome: Change From Baseline in Mean Intra Ocular Pressure (IOP) in Study Eye at Day 15: 4 AM (20 Hours)
Description: IOP was measured using Perkins applanation tonometer at Day -8 and using standard Goldmann applanation tonometer at eligibility visit, Day -7 and Day 15. IOP was measured in both eyes, and the eye with higher IOP reading across eligibility visit and Day -8 was referred as 'study eye' for efficacy assessment. If both measurements were equal, right eye was selected as study eye. IOP was measured twice in the same eye, and if difference between 2 measurements was less than or equal to 2 millimeter of mercury (mmHg), mean of 2 readings was recorded as IOP at that time point. If the difference between 2 readings was greater than 2 mmHg, a third consecutive reading was taken and the median IOP was recorded as the IOP at that time point. Mean IOP was reported as the average of individual participants' mean or median IOP values. Change from baseline in IOP = baseline IOP - post-baseline IOP. Change was calculated using the value at 4 AM on Day -7 as baseline for 4 AM value on Day 15.
Time Frame: 4 AM on Baseline (Day -7), 4 AM on Day 15 (20 Hours)
Population: PP population included all participants who completed the study treatment with no major protocol violations.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Taprenepag+Latanoprost | Taprenepag+Latanoprost Vehicle
Number analyzed (Participants) | 24 | 28
mmHg
  Baseline (Day -7) : 4 AM | 16.77 (3.742) | 16.66 (2.941)
  Change at Day 15: 4 AM | 4.31 (3.978) | 4.39 (2.551)

11. Primary Outcome: Change From Baseline in Mean Intra Ocular Pressure (IOP) in Study Eye at Day 15: 6 AM (22 Hours)
Description: IOP was measured using Perkins applanation tonometer at Day -8 and using standard Goldmann applanation tonometer at eligibility visit, Day -7 and Day 15. IOP was measured in both eyes, and the eye with higher IOP reading across eligibility visit and Day -8 was referred as 'study eye' for efficacy assessment. If both measurements were equal, right eye was selected as study eye. IOP was measured twice in the same eye, and if difference between 2 measurements was less than or equal to 2 millimeter of mercury (mmHg), mean of 2 readings was recorded as the IOP at that time point. If difference between 2 readings was greater than 2 mmHg, a third consecutive reading was taken and the median IOP was recorded as the IOP at that time point. Mean IOP was reported as the average of individual participants' mean or median IOP values. Change from baseline in IOP = baseline IOP - post-baseline IOP. Change was calculated using the value at 6 AM on Day -7 as baseline for 6 AM value on Day 15.
Time Frame: 6 AM on Baseline (Day -7), 6 AM on Day 15 (22 Hours)
Population: PP population included all participants who completed the study treatment with no major protocol violations.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Taprenepag+Latanoprost | Taprenepag+Latanoprost Vehicle
Number analyzed (Participants) | 24 | 28
mmHg
  Baseline (Day -7): 6 AM | 17.98 (3.952) | 17.36 (2.785)
  Change at Day 15: 6 AM | 5.02 (4.415) | 4.32 (2.878)

12. Primary Outcome: Change From Baseline in Mean Intra Ocular Pressure (IOP) in Study Eye at Day 15: 8 AM (24 Hours)
Description: IOP was measured using Perkins applanation tonometer at Day -8 and using standard Goldmann applanation tonometer at eligibility visit, Day -7 and Day 15. IOP was measured in both eyes, and the eye with higher IOP reading across eligibility visit and Day -8 was referred as 'study eye' for efficacy assessment. If both measurements were equal, right eye was selected as study eye. IOP was measured twice in the same eye, and if difference between 2 measurements was less than or equal to 2 millimeter of mercury (mmHg), mean of 2 readings was recorded as IOP at that time point. If the difference between 2 readings was greater than 2 mmHg, a third consecutive reading was taken and the median IOP was recorded as the IOP at that time point. Mean IOP was reported as the average of individual participants' mean or median IOP values. Change from baseline in IOP = baseline IOP - post-baseline IOP. Change was calculated using the value at 8 AM on Day -7 as baseline for 8 AM value on Day 15.
Time Frame: 8 AM on Baseline (Day -7), 8 AM on Day 15 (24 Hours)
Population: PP population included all participants who completed the study treatment with no major protocol violations.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Taprenepag+Latanoprost | Taprenepag+Latanoprost Vehicle
Number analyzed (Participants) | 24 | 28
mmHg
  Baseline (Day -7): 8 AM | 23.31 (2.497) | 22.71 (2.347)
  Change at Day 15: 8 AM | 6.19 (2.801) | 4.77 (2.518)

13. Primary Outcome: Change From Baseline in Mean Intra Ocular Pressure (IOP) in Study Eye at Day 16: 8 AM (48 Hours)
Description: IOP was measured using Perkins applanation tonometer at Day -8 and using standard Goldmann applanation tonometer at eligibility visit and Day 16. IOP was measured in both eyes, and the eye with higher IOP reading across eligibility visit and Day -8 was referred as 'study eye' for efficacy assessment. If both measurements were equal, right eye was selected as study eye. IOP was measured twice in the same eye, and if difference between 2 measurements was less than or equal to 2 millimeter of mercury (mmHg), the mean of 2 readings was recorded as the IOP at that time point. If the difference between 2 readings was greater than 2 mmHg, a third consecutive reading was taken and the median IOP was recorded as the IOP at that time point. Mean IOP was reported as the average of individual participants' mean or median IOP values. Change from baseline in IOP = baseline IOP - post-baseline IOP. Change was calculated using the value at 8 AM on Day -8 as baseline for 8 AM value on Day 16.
Time Frame: 8 AM on Baseline (Day -8), 8 AM on Day 16 (48 Hours)
Population: PP population included all participants who completed the study treatment with no major protocol violations.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Taprenepag+Latanoprost | Taprenepag+Latanoprost Vehicle
Number analyzed (Participants) | 24 | 28
mmHg | 1.21 (5.009) | -0.20 (3.023)

14. Primary Outcome: Change From Baseline in Mean Intra Ocular Pressure (IOP) in Study Eye at Day 17: 8 AM (72 Hours)
Description: IOP was measured using Perkins applanation tonometer at Day -8 and using standard Goldmann applanation tonometer at eligibility visit and Day 17. IOP was measured in both eyes, and the eye with higher IOP reading across eligibility visit and Day -8 was referred as 'study eye' for efficacy assessment. If both measurements were equal, right eye was selected as study eye. IOP was measured twice in the same eye, and if difference between 2 measurements was less than or equal to 2 millimeter of mercury (mmHg), the mean of 2 readings was recorded as the IOP at that time point. If the difference between 2 readings was greater than 2 mmHg, a third consecutive reading was taken and the median IOP was recorded as the IOP at that time point. Mean IOP was reported as the average of individual participants' mean or median IOP values. Change from baseline in IOP = baseline IOP - post-baseline IOP. Change was calculated using the value at 8 AM on Day -8 as baseline for 8 AM value on Day 17.
Time Frame: 8 AM on Baseline (Day -8), 8 AM on Day 17 (72 Hours)
Population: PP population included all participants who completed the study treatment with no major protocol violations. Here 'overall number of participants analyzed) signifies those participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Taprenepag+Latanoprost | Taprenepag+Latanoprost Vehicle
Number analyzed (Participants) | 23 | 28
mmHg | 0.89 (3.769) | -0.95 (3.563)

15. Primary Outcome: Change From Baseline in Mean Intra Ocular Pressure (IOP) in Study Eye at Day 21: 8 AM (168 Hours)
Description: IOP was measured using Perkins applanation tonometer at Day -8 and using standard Goldmann applanation tonometer at eligibility visit and Day 21. IOP was measured in both eyes, and the eye with higher IOP reading across eligibility visit and Day -8 was referred as 'study eye' for efficacy assessment. If both measurements were equal, right eye was selected as study eye. IOP was measured twice in the same eye, and if difference between 2 measurements was less than or equal to 2 millimeter of mercury (mmHg), the mean of 2 readings was recorded as the IOP at that time point. If the difference between 2 readings was greater than 2 mmHg, a third consecutive reading was taken and the median IOP was recorded as the IOP at that time point. Mean IOP was reported as the average of individual participants' mean or median IOP values. Change from baseline in IOP = baseline IOP - post-baseline IOP. Change was calculated using the value at 8 AM on Day -8 as baseline for 8 AM value on Day 21.
Time Frame: 8 AM on Day -8 (Baseline), 8 AM on Day 21 (168 Hours)
Population: PP population included all participants who completed the study treatment with no major protocol violations.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Taprenepag+Latanoprost | Taprenepag+Latanoprost Vehicle
Number analyzed (Participants) | 24 | 28
mmHg | -0.19 (3.017) | -0.36 (3.197)

16. Primary Outcome: Plasma Concentration for PF-04217329 Active Metabolite (CP-544326) at 5 Minutes on Day 14
Time Frame: 5 minutes post-dose on Day 14
Population: Evaluable PK population included all enrolled participants who completed study treatment, had at least 1 quantifiable concentration (that is, at least 1 concentration above the limit of quantification) and had no major protocol deviation. Here 'overall number of participants analyzed' signifies those participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Taprenepag+Latanoprost | Taprenepag+Latanoprost Vehicle
Number analyzed (Participants) | 26 | 27
pg/mL | 36.20 (23.847) | 43.27 (36.290)

17. Primary Outcome: Plasma Concentration for PF-04217329 Active Metabolite (CP-544326) at 0.25 Hours on Day 14
Time Frame: 0.25 hours post-dose on Day 14
Population: Evaluable PK population included all enrolled participants who completed study treatment, had at least 1 quantifiable concentration (that is, at least 1 concentration above the limit of quantification) and had no major protocol deviation.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Taprenepag+Latanoprost | Taprenepag+Latanoprost Vehicle
Number analyzed (Participants) | 26 | 28
pg/mL | 67.23 (33.885) | 88.65 (54.679)

18. Primary Outcome: Plasma Concentration for PF-04217329 Active Metabolite (CP-544326) at 0.5 Hours on Day 14
Time Frame: 0.5 hours post-dose on Day 14
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Taprenepag+Latanoprost | Taprenepag+Latanoprost Vehicle
Number analyzed (Participants) | 26 | 28
pg/mL | 47.88 (29.811) | 53.07 (34.336)

19. Primary Outcome: Plasma Concentration for PF-04217329 Active Metabolite (CP-544326) at 0.75 Hours on Day 14
Time Frame: 0.75 hours post-dose on Day 14
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Taprenepag+Latanoprost | Taprenepag+Latanoprost Vehicle
Number analyzed (Participants) | 26 | 28
pg/mL | 31.68 (20.692) | 30.74 (18.726)

20. Primary Outcome: Plasma Concentration for PF-04217329 Active Metabolite (CP-544326) at 1 Hour on Day 14
Time Frame: 1 hour post-dose on Day 14
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Taprenepag+Latanoprost | Taprenepag+Latanoprost Vehicle
Number analyzed (Participants) | 26 | 28
pg/mL | 24.94 (25.301) | 18.96 (14.827)

21. Secondary Outcome: Diastolic Ocular Perfusion Pressure (DOPP)
Description: DOPP = diastolic blood pressure minus IOP of the study eye. IOP was measured using Perkins applanation tonometer at Day -8, Day 14 and using standard Goldmann applanation tonometer at eligibility visit and Day 15. IOP was measured in both the eyes, and the eye with higher IOP reading across eligibility visit and Day -8 was referred as 'study eye' for efficacy assessment. If both the measurements were equal, right eye was selected as the study eye.
Time Frame: 8 AM, 10 AM, 12 PM, 2 PM, 4 PM, 6 PM, 8 PM, 10 PM on Day 14; 12 AM, 4 AM, 6 AM, 8 AM on Day 15
Population: The intent-to-treat population included all randomized participants who receive at least 1 dose of study medication. Here 'number analyzed' signifies those participants who were evaluable for this measure at given time points for each group, respectively. Last observation carried forward (LOCF) was used to impute missing data.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Taprenepag+Latanoprost | Taprenepag+Latanoprost Vehicle
Number analyzed (Participants) | 30 | 29
mmHg
  Day 14: 8AM | 57.42 (8.984) | 57.48 (12.100)
  Day 14: 10AM | 48.28 (10.902) | 48.29 (10.652)
  Day 14: 12PM | 52.70 (10.289) | 52.84 (10.105)
  Day 14: 2PM: number analyzed (Participants) | 30 | 28
  Day 14: 2PM | 49.73 (12.744) | 52.52 (10.908)
  Day 14: 4PM: number analyzed (Participants) | 30 | 28
  Day 14: 4PM | 56.73 (9.555) | 56.75 (9.776)
  Day 14: 6PM | 59.38 (9.527) | 60.41 (9.809)
  Day 14: 8PM | 58.18 (10.929) | 55.98 (10.351)
  Day 14: 10PM | 51.57 (12.317) | 49.86 (10.419)
  Day 15: 12AM | 51.10 (10.247) | 53.52 (12.302)
  Day 15: 4AM | 54.25 (11.929) | 54.00 (11.168)
  Day 15: 6AM | 54.08 (11.784) | 53.90 (11.385)
  Day 15: 8AM | 57.32 (10.431) | 58.47 (10.941)

22. Secondary Outcome: Change From Baseline in Diastolic Ocular Perfusion Pressure (DOPP) at Day 14 (8 AM, 10 AM, 12 PM, 2 PM, 4 PM, 6 PM, 8 PM, 10 PM) and Day 15 (12 AM, 2 AM, 4 AM, 6 AM and 8 AM)
Description: DOPP=diastolic blood pressure minus IOP of the study eye. IOP was measured using Perkins applanation tonometer at Day -8, Day 14 and using standard Goldmann applanation tonometer at eligibility visit, Day -7 and Day 15. IOP was measured in both the eyes, and the eye with higher IOP reading across eligibility visit and Day -8 was referred as 'study eye' for efficacy assessment. If both the measurements were equal, right eye was selected as the study eye. Change at various post-dose time points on Day 14 and Day 15 was calculated from the values at same time points on Day -8 and Day -7 respectively (for example, value at 8 AM on Day -8 was used as baseline value for 8 AM value on Day 14 and value at 8 AM on Day -7 was used as baseline value for 8 AM value on Day 15).
Time Frame: 8 AM, 10 AM, 12 PM, 2 PM, 4 PM, 6 PM, 8 PM, and 10 PM on Day -8 (Baseline), Day 14; 12 AM, 4 AM, 6 AM, 8 AM on Day -7 (Baseline), Day 15
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Taprenepag+Latanoprost | Taprenepag+Latanoprost Vehicle
Number analyzed (Participants) | 24 | 28
mmHg
  Day -8: Baseline for Day 14 8 AM (n=24,28) | 52.81 (11.179) | 53.05 (13.183)
  Day -8: Baseline for Day 14 10 AM(n=24,28) | 46.06 (10.862) | 44.57 (13.493)
  Day -8: Baseline for Day 14 12 PM (n=24,28) | 47.29 (10.917) | 50.34 (11.341)
  Day -8: Baseline for Day 14 2 PM (n=24,28) | 46.75 (10.260) | 46.13 (9.988)
  Day -8: Baseline for Day 14 4 PM (n=24,28) | 53.98 (13.218) | 52.39 (10.495)
  Day -8: Baseline for Day 14 6 PM (n=24,28) | 53.98 (12.883) | 58.14 (12.280)
  Day -8: Baseline for Day 14 8 PM (n=24,28) | 52.50 (15.829) | 53.77 (13.349)
  Day -8: Baseline for Day 14 10 PM (n=24,28) | 46.54 (9.894) | 47.79 (14.196)
  Day -7: Baseline for Day 15 12 AM (n=24,28) | 48.73 (9.880) | 49.73 (11.843)
  Day -7: Baseline for Day 15 4 AM (n=24,28) | 51.98 (12.386) | 51.73 (10.801)
  Day -7: Baseline for Day 15: 6 AM | 53.60 (13.672) | 54.39 (13.151)
  Day -7: Baseline for Day 15: 8 AM | 52.94 (10.584) | 55.18 (11.923)
  Change at Day 14: 8 AM | 5.38 (8.403) | 4.43 (7.262)
  Change at Day 14: 10 AM | 2.77 (9.336) | 3.70 (11.108)
  Change at Day 14: 12 PM | 6.65 (8.906) | 2.82 (8.790)
  Change at Day 14: 2 PM: number analyzed (Participants) | 24 | 27
  Change at Day 14: 2 PM | 4.15 (12.645) | 7.31 (7.558)
  Change at Day 14: 4 PM: number analyzed (Participants) | 24 | 27
  Change at Day 14: 4 PM | 3.25 (13.492) | 3.98 (7.597)
  Change at Day 14: 6 PM | 6.00 (10.208) | 2.59 (10.723)
  Change at Day 14: 8 PM | 6.94 (11.900) | 2.16 (8.423)
  Change at Day 14: 10 PM | 5.73 (10.332) | 2.05 (10.401)
  Change at Day 15: 12 AM | 3.04 (6.716) | 3.80 (8.231)
  Change at Day 15: 4 AM | 2.85 (8.222) | 1.86 (6.592)
  Change at Day 15: 6 AM | 1.81 (8.899) | -0.43 (7.595)
  Change at Day 15: 8 AM | 4.23 (8.180) | 3.23 (9.857)
Statistical Analysis 1: Comparison: Taprenepag+Latanoprost vs Taprenepag+Latanoprost Vehicle; Change at Day 14 8 AM: Analysis was based on analysis of covariance (ANCOVA) using statistical analysis system (SAS) mixed procedure with covariates of baseline IOP, sequence, study period and treatment as fixed effects and participant within sequence as random effect; Test type: Superiority or Other; p = 0.5330, ANCOVA; Mean Difference (Final Values) = 1.07, 90% CI 2-sided [-1.82 to 3.95]
Statistical Analysis 2: Comparison: Taprenepag+Latanoprost vs Taprenepag+Latanoprost Vehicle; Change at Day 14 10 AM: Analysis was based on ANCOVA using SAS mixed procedure with covariates of baseline IOP, sequence, study period and treatment as fixed effects and participant within sequence as random effect; Test type: Superiority or Other; p = 0.9532, ANCOVA; Mean Difference (Final Values) = -0.14, 90% CI 2-sided [-4.13 to 3.85]
Statistical Analysis 3: Comparison: Taprenepag+Latanoprost vs Taprenepag+Latanoprost Vehicle; Change at Day 14 12 PM: Analysis was based on ANCOVA using SAS mixed procedure with covariates of baseline IOP, sequence, study period and treatment as fixed effects and participant within sequence as random effect; Test type: Superiority or Other; p = 0.2493, ANCOVA; Mean Difference (Final Values) = 2.53, 90% CI 2-sided [-1.11 to 6.18]
Statistical Analysis 4: Comparison: Taprenepag+Latanoprost vs Taprenepag+Latanoprost Vehicle; Change at Day 14 2 PM: Analysis was based on ANCOVA using SAS mixed procedure with covariates of baseline IOP, sequence, study period and treatment as fixed effects and participant within sequence as random effect; Test type: Superiority or Other; p = 0.2801, ANCOVA; Mean Difference (Final Values) = -2.99, 90% CI 2-sided [-7.59 to 1.60]
Statistical Analysis 5: Comparison: Taprenepag+Latanoprost vs Taprenepag+Latanoprost Vehicle; Change at Day 14 4 PM: Analysis was based on ANCOVA using SAS mixed procedure with covariates of baseline IOP, sequence, study period and treatment as fixed effects and participant within sequence as random effect; Test type: Superiority or Other; p = 0.9288, ANCOVA; Mean Difference (Final Values) = -0.19, 90% CI 2-sided [-3.77 to 3.39]
Statistical Analysis 6: Comparison: Taprenepag+Latanoprost vs Taprenepag+Latanoprost Vehicle; Change at Day 14 6 PM: Analysis was based on ANCOVA using SAS mixed procedure with covariates of baseline IOP, sequence, study period and treatment as fixed effects and participant within sequence as random effect; Test type: Superiority or Other; p = 0.6459, ANCOVA; Mean Difference (Final Values) = 0.98, 90% CI 2-sided [-2.62 to 4.58]
Statistical Analysis 7: Comparison: Taprenepag+Latanoprost vs Taprenepag+Latanoprost Vehicle; Change at Day 14 8 PM: Analysis was based on ANCOVA using SAS mixed procedure with covariates of baseline IOP, sequence, study period and treatment as fixed effects and participant within sequence as random effect; Test type: Superiority or Other; p = 0.0527, ANCOVA; Mean Difference (Final Values) = 4.06, 90% CI 2-sided [0.63 to 7.48]
Statistical Analysis 8: Comparison: Taprenepag+Latanoprost vs Taprenepag+Latanoprost Vehicle; Change at Day 14 10 PM: Analysis was based on ANCOVA using SAS mixed procedure with covariates of baseline IOP, sequence, study period and treatment as fixed effects and participant within sequence as random effect; Test type: Superiority or Other; p = 0.1998, ANCOVA; Mean Difference (Final Values) = 3.29, 90% CI 2-sided [-0.95 to 7.52]
Statistical Analysis 9: Comparison: Taprenepag+Latanoprost vs Taprenepag+Latanoprost Vehicle; Change at Day 15 12 AM: Analysis was based on ANCOVA using SAS mixed procedure with covariates of baseline IOP, sequence, study period and treatment as fixed effects and participant within sequence as random effect; Test type: Superiority or Other; p = 0.6765, ANCOVA; Mean Difference (Final Values) = -0.85, 90% CI 2-sided [-4.22 to 2.53]
Statistical Analysis 10: Comparison: Taprenepag+Latanoprost vs Taprenepag+Latanoprost Vehicle; Change at Day 15 4 AM: Analysis was based on ANCOVA using SAS mixed procedure with covariates of baseline IOP, sequence, study period and treatment as fixed effects and participant within sequence as random effect; Test type: Superiority or Other; p = 0.6221, ANCOVA; Mean Difference (Final Values) = 0.99, 90% CI 2-sided [-2.35 to 4.33]
Statistical Analysis 11: Comparison: Taprenepag+Latanoprost vs Taprenepag+Latanoprost Vehicle; Change at Day 15 6 AM: Analysis was based on ANCOVA using SAS mixed procedure with covariates of baseline IOP, sequence, study period and treatment as fixed effects and participant within sequence as random effect; Test type: Superiority or Other; p = 0.3000, ANCOVA; Mean Difference (Final Values) = 1.81, 90% CI 2-sided [-1.11 to 4.74]
Statistical Analysis 12: Comparison: Taprenepag+Latanoprost vs Taprenepag+Latanoprost Vehicle; Change at Day 15 8 AM: Analysis was based on ANCOVA using SAS mixed procedure with covariates of baseline IOP, sequence, study period and treatment as fixed effects and participant within sequence as random effect; Test type: Superiority or Other; p = 0.9103, ANCOVA; Mean Difference (Final Values) = -0.24, 90% CI 2-sided [-3.85 to 3.37]

23. Secondary Outcome: Number of Participants With Ocular and Systemic Adverse Events (AEs)
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. Treatment-emergent are events between first dose of study medication and up to 28 days after last dose that were absent before treatment or that worsened relative to pretreatment state. Number of participants with ocular (AE related to eye) and systemic (all AEs including eye) AEs were reported.
Time Frame: Baseline up to 28 days after last dose of study medication (up to 58 Days)
Population: Intent-to-treat (ITT) population included all randomized participants who received at least 1 dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Taprenepag+Latanoprost | Taprenepag+Latanoprost Vehicle
Number analyzed (Participants) | 30 | 29
Participants
  Ocular AEs | 29 | 25
  Systemic AEs | 30 | 28

24. Secondary Outcome: Percentage of Participants With Photophobia and Iritis
Description: Percentage of participants with treatment emergent photophobia (abnormal sensitivity or intolerance of eye towards light) and iritis (inflammation of the iris of eye) were reported. Treatment-emergent are events between first dose of study medication and up to 28 days after last dose that were absent before treatment or that worsened relative to pretreatment state.
Time Frame: Baseline up to 28 days after last dose of study medication (up to 58 Days)
Population: ITT population included all randomized participants who received at least 1 dose of study medication.
Measure: Number; unit: percentage of participants
Arm/Group | Taprenepag+Latanoprost | Taprenepag+Latanoprost Vehicle
Number analyzed (Participants) | 30 | 29
percentage of participants
  Photophobia | 83.33 | 24.14
  Iritis | 3.33 | 6.90
Statistical Analysis 1: Comparison: Taprenepag+Latanoprost vs Taprenepag+Latanoprost Vehicle; Photophobia: p-value was calculated using fisher exact test; Test type: Superiority or Other; p < 0.001, Fisher Exact; Percent Difference = 59.20, 95% CI 2-sided [38.69 to 79.70]
Statistical Analysis 2: Comparison: Taprenepag+Latanoprost vs Taprenepag+Latanoprost Vehicle; Iritis: p-value was calculated using fisher exact test; Test type: Superiority or Other; p = 0.612, Fisher Exact; Percent Difference = -3.56, 95% CI 2-sided [-14.80 to 7.68]

25. Secondary Outcome: Change From Baseline in Corneal Thickness at Day 7, 13, 16, 21, 28 and 35
Description: Corneal thickness was measured using an ultrasonic pachymeter. Corneal thickness in both study eye and fellow eye were reported. Study eye: IOP was measured in both the eyes, and the eye with higher IOP reading across eligibility visit and Day -8 was referred as 'study eye'. If both the measurements were equal, right eye was selected as the study eye. The other eye was referred as 'fellow eye'.
Time Frame: 8 AM on Day 1 (Baseline), Days 7, 13, 16, 21, 28, 35
Population: ITT population included all randomized participants who received at least 1 dose of study medication.
Measure: Mean (Standard Deviation); unit: micrometer
Arm/Group | Taprenepag+Latanoprost | Taprenepag+Latanoprost Vehicle
Number analyzed (Participants) | 30 | 29
micrometer
  Day 1 8 AM: Baseline for study eye | 562.8 (24.11) | 561.0 (25.94)
  Day 1 8 AM: Baseline for fellow eye | 562.5 (24.86) | 560.7 (28.36)
  Change at Day 7 8 AM: study eye | 26.6 (21.55) | 25.0 (16.20)
  Change at Day 7 8 AM: fellow eye | 26.7 (19.81) | 26.4 (18.12)
  Change at Day 13 8 AM: study eye | 20.2 (22.86) | 21.2 (16.35)
  Change at Day 13 8 AM: fellow eye | 24.4 (19.63) | 24.9 (20.42)
  Change at Day 16 8 AM: study eye | 20.7 (16.70) | 19.7 (17.93)
  Change at Day 16 8 AM: fellow eye | 21.7 (18.77) | 22.0 (18.41)
  Change at Day 21 8 AM: study eye | 5.7 (13.00) | 8.9 (10.42)
  Change at Day 21 8 AM: fellow eye | 6.4 (10.09) | 10.9 (13.38)
  Change at Day 28 8 AM: study eye | 7.8 (15.93) | 6.9 (11.69)
  Change at Day 28 8 AM: fellow eye | 8.2 (9.20) | 9.2 (9.88)
  Change at Day 35 8 AM: study eye | 2.3 (13.20) | 5.4 (10.60)
  Change at Day 35 8 AM: fellow eye | 5.1 (10.99) | 5.9 (12.79)

26. Secondary Outcome: Change From Baseline in Corneal Endothelial Cell Counts at Day 13 and 35
Description: Endothelial cell count was defined as the number of cells per millimeter square (cells/mm^2) of endothelium and was calculated using confocal microscopy for both study eye and fellow eye. Study eye: IOP was measured in both the eyes, and the eye with higher IOP reading across eligibility visit and Day -8 was referred as 'study eye'. If both the measurements were equal, right eye was selected as the study eye. The other eye was referred as 'fellow eye'.
Time Frame: 8 AM on Day 1 (Baseline), Day 13, 35
Population: ITT population included all randomized participants who received at least 1 dose of study medication. Here 'number analyzed' signifies those participants who were evaluable for this outcome measure at given time points, for each group respectively.
Measure: Mean (Standard Deviation); unit: cells/mm^2
Arm/Group | Taprenepag+Latanoprost | Taprenepag+Latanoprost Vehicle
Number analyzed (Participants) | 30 | 29
cells/mm^2
  Day 1 8 AM: Baseline for study eye: number analyzed (Participants) | 30 | 28
  Day 1 8 AM: Baseline for study eye | 2560.7 (501.79) | 2585.3 (460.49)
  Day 1 8 AM: Baseline for fellow eye | 2456.5 (476.69) | 2519.1 (440.66)
  Change at Day 13 8 AM: study eye: number analyzed (Participants) | 30 | 28
  Change at Day 13 8 AM: study eye | -41.8 (162.76) | 17.2 (192.40)
  Change at Day 13 8 AM: fellow eye | 29.5 (127.07) | -12.1 (130.47)
  Change at Day 35 8 AM: study eye: number analyzed (Participants) | 29 | 28
  Change at Day 35 8 AM: study eye | -10.6 (140.50) | -45.3 (136.64)
  Change at Day 35 8 AM: fellow eye: number analyzed (Participants) | 29 | 29
  Change at Day 35 8 AM: fellow eye | -12.6 (147.25) | -13.4 (122.50)
Statistical Analysis 1: Comparison: Taprenepag+Latanoprost vs Taprenepag+Latanoprost Vehicle; Change at Day 13 8 AM study eye: Analysis was based on ANCOVA using SAS mixed procedure with covariates of baseline IOP, sequence, study period and treatment as fixed effects and participant within sequence as random effect; Test type: Superiority or Other; p = 0.2450, ANCOVA; Mean Difference (Final Values) = -52.42, 90% CI 2-sided [-127.05 to 22.22]
Statistical Analysis 2: Comparison: Taprenepag+Latanoprost vs Taprenepag+Latanoprost Vehicle; Change at Day 13 8 AM fellow eye: Analysis was based on ANCOVA using SAS mixed procedure with covariates of baseline IOP, sequence, study period and treatment as fixed effects and participant within sequence as random effect; Test type: Superiority or Other; p = 0.3068, ANCOVA; Mean Difference (Final Values) = 34.51, 90% CI 2-sided [-21.89 to 90.91]
Statistical Analysis 3: Comparison: Taprenepag+Latanoprost vs Taprenepag+Latanoprost Vehicle; Change at Day 35 8 AM study eye: Analysis was based on ANCOVA using SAS mixed procedure with covariates of baseline IOP, sequence, study period and treatment as fixed effects and participant within sequence as random effect; Test type: Superiority or Other; p = 0.2632, ANCOVA; Mean Difference (Final Values) = 40.99, 90% CI 2-sided [-19.69 to 101.67]
Statistical Analysis 4: Comparison: Taprenepag+Latanoprost vs Taprenepag+Latanoprost Vehicle; Change at Day 35 8 AM fellow eye: Analysis was based on ANCOVA using SAS mixed procedure with covariates of baseline IOP, sequence, study period and treatment as fixed effects and participant within sequence as random effect; Test type: Superiority or Other; p = 0.8373, ANCOVA; Mean Difference (Final Values) = -6.60, 90% CI 2-sided [-60.84 to 47.64]

27. Other Pre Specified Outcome: Maximum Conjunctival Hyperemia Score
Description: Conjunctival hyperemia score was assessed using slit-lamp examination on a photographic reference scale ranging from 0 (normal) to 3 (severe). Higher score indicated severe condition. Conjunctival hyperemia was recorded to the nearest whole number using standard rounding rules (for example, a score of 1.5 was rounded up to 2 and a score of 1.4 was rounded down to 1). Highest conjunctival hyperemia score observed at Day -8 (baseline) and through Day 1 to 35 were reported. Maximum conjunctival hyperemia score for both study eye and fellow eye was reported. Study eye: IOP was measured in both the eyes, and the eye with higher IOP reading across eligibility visit and Day -8 was referred as 'study eye'. If both the measurements were equal, right eye was selected as the study eye. The other eye was referred as 'fellow eye'.
Time Frame: Day -8 (Baseline), Day 1 to 35
Population: ITT population included all randomized participants who received at least 1 dose of study medication.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Taprenepag+Latanoprost | Taprenepag+Latanoprost Vehicle
Number analyzed (Participants) | 30 | 29
units on a scale
  Day -8: Baseline for study eye | 0.30 (0.466) | 0.38 (0.494)
  Day -8: Baseline for fellow eye | 0.30 (0.466) | 0.28 (0.455)
  Day 1 to 35: study eye | 1.87 (0.776) | 1.45 (0.632)
  Day 1 to 35: fellow eye | 1.77 (0.898) | 1.38 (0.728)

28. Other Pre Specified Outcome: Change From Baseline in Maximum Conjunctival Hyperemia Score Observed
Description: Conjunctival hyperemia score was assessed using slit-lamp examination on a photographic reference scale ranging from 0 (normal) to 3 (severe). Conjunctival hyperemia was recorded to the nearest whole number using standard rounding rules (for example, a score of 1.5 was rounded up to 2 and a score of 1.4 was rounded down to 1). Change between highest conjunctival hyperemia score observed through Day 1 to 35 and highest conjunctival hyperemia score at baseline (Day -8) was reported. Maximum conjunctival hyperemia score for both study eye and fellow eye was reported. Study eye: IOP was measured in both the eyes, and the eye with higher IOP reading across eligibility visit and Day -8 was referred as 'study eye'. If both the measurements were equal, right eye was selected as the study eye. The other eye was referred as 'fellow eye'.
Time Frame: Day -8 (Baseline), Day 1 to 35
Population: ITT population included all randomized participants who received at least 1 dose of study medication.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Taprenepag+Latanoprost | Taprenepag+Latanoprost Vehicle
Number analyzed (Participants) | 30 | 29
units on a scale
  Change in study eye | 1.57 (0.679) | 1.07 (0.593)
  Change in fellow eye | 1.47 (0.860) | 1.10 (0.673)

29. Other Pre Specified Outcome: Total Corneal Staining Score
Description: Corneal staining was assessed using fluorescein dye, a yellow filter, and a slit lamp. The cornea was divided into 5 different zones. Each corneal zone was graded independently using a 0 to 3 grading scale; where 0= no staining, 1= scattered micropunctate staining (dots were discrete and countable), 2= areas of clustered micropunctate or one macropunctate stain, 3= areas of confluent micropunctate stain or two or more macropunctate stain or filaments. Sum of scores of each zone led to total score. Total score range: 0 to 15, higher score indicated greater staining. Total corneal score from both study eye and fellow eye were reported. Study eye: IOP was measured in both the eyes, and the eye with higher IOP reading across eligibility visit and baseline visit was referred as 'study eye'. If both the measurements were equal, right eye was selected as the study eye. The other eye was referred as 'fellow eye'.
Time Frame: 8 AM on Day 1 (Baseline)
Population: ITT population included all randomized participants who received at least 1 dose of study medication.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Taprenepag+Latanoprost | Taprenepag+Latanoprost Vehicle
Number analyzed (Participants) | 30 | 29
units on a scale
  Day 1 8 AM: Baseline for study eye | 0.1 (0.25) | 0.0 (0.00)
  Day 1 8 AM: Baseline for fellow eye | 0.0 (0.18) | 0.0 (0.00)

30. Other Pre Specified Outcome: Change From Baseline in Total Corneal Staining Score at Day 7, 13, 16, 21, 28 and 35
Description: as for outcome 29
Time Frame: 8 AM Day 1 (Baseline), Day 7, 13, 16, 21, 28, 35
Population: ITT population included all randomized participants who received at least 1 dose of study medication.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Taprenepag+Latanoprost | Taprenepag+Latanoprost Vehicle
Number analyzed (Participants) | 30 | 29
units on a scale
  Change at Day 7 8 AM: study eye | 0.6 (1.28) | 0.3 (0.81)
  Change at Day 7 8 AM: fellow eye | 0.5 (0.90) | 0.4 (0.87)
  Change at Day 13 8 AM: study eye | 0.9 (1.44) | 1.0 (1.48)
  Change at Day 13 8 AM: fellow eye | 0.9 (1.67) | 1.0 (1.74)
  Change at Day 16 8 AM: study eye | 0.7 (1.49) | 1.1 (1.48)
  Change at Day 16 8 AM: fellow eye | 0.8 (1.56) | 0.9 (1.40)
  Change at Day 21 8 AM: study eye | 0.4 (0.81) | 0.4 (0.90)
  Change at Day 21 8 AM: fellow eye | 0.4 (0.86) | 0.2 (0.69)
  Change at Day 28 8 AM: study eye | 0.1 (0.61) | 0.3 (0.65)
  Change at Day 28 8 AM: fellow eye | 0.1 (0.45) | 0.0 (0.00)
  Change at Day 35 8 AM: study eye | -0.0 (0.32) | 0.0 (0.19)
  Change at Day 35 8 AM: fellow eye | -0.0 (0.18) | 0.0 (0.00)

ADVERSE EVENTS:
Time Frame: Baseline up to 28 days after last dose of study medication (up to 58 Days)
Description: ITT population, which included all randomized participants who received at least 1 dose of study medication.
Arm/Group | Taprenepag+Latanoprost | Taprenepag+Latanoprost Vehicle
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/29
Other Adverse Events (participants affected / at risk) | 30/30 | 28/29
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Taprenepag+Latanoprost (N=30) | Taprenepag+Latanoprost Vehicle (N=29)
Asthenopia (Eye disorders) | 1 | 0
Conjunctival hyperaemia (Eye disorders) | 13 | 13
Corneal disorder (Eye disorders) | 23 | 22
Dry eye (Eye disorders) | 1 | 2
Eye pain (Eye disorders) | 5 | 1
Eye pruritus (Eye disorders) | 1 | 0
Iritis (Eye disorders) | 1 | 2
Lacrimation increased (Eye disorders) | 0 | 1
Ocular hyperaemia (Eye disorders) | 2 | 0
Photophobia (Eye disorders) | 25 | 7
Vision blurred (Eye disorders) | 3 | 3
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Instillation site pain (General disorders) | 2 | 1
Sensation of foreign body (General disorders) | 2 | 0
Food allergy (Immune system disorders) | 1 | 0
Fungal infection (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 3 | 3
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 1 | 0
Blood potassium increased (Investigations) | 1 | 1
Corneal staining (Investigations) | 20 | 20
Costochondritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Headache (Nervous system disorders) | 6 | 5
Sciatica (Nervous system disorders) | 1 | 1
Uterine prolapse (Reproductive system and breast disorders) | 1 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.